CLINICAL TRIAL: NCT06477627
Title: The Coastal Exposome: a Study of Sea Air Inhalation and Possible Links to Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0078
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Immune Suppression; Exposure
Keywords: Oceans and human health

STUDY DESIGN:
Intervention Model Description: three groups: one group that lives at the coast all year round, one group that lives inland all year round and one group that live inland but in the month August lives at the coast (to investigate the change in environment) The participants will not get any treatment, they just have to give samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Studygroup that will move from inland to the coast for one month (Other): This group normally lives inland and live at the coast in august. We investigate the change to the coast environment
  Interventions: Other: change of environment
- reference group coast (Other): This group lives inland the whole year round
  Interventions: Other: no intervention
- reference group inland (Other): This group lives inland all year round.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: change of environment — The participants will change from inland to coastal environment to see the effect. We will take VAMS blood samples and nose swabs from the participant to measure this effect.
  Arms: Studygroup that will move from inland to the coast for one month
Other: no intervention — reference groups, stay in their coastal or inland environment
  Arms: reference group coast; reference group inland

SUMMARY:
The research aims to understand oceans as crucial contributors to human health in coastal environments. Oceans produce marine spray aerosols that contain a mixture of microbiota and natural biological molecules (biogenics).

DETAILED DESCRIPTION:
The primary outcome envisioned consists of 2 goals.

1. In this study, the first objective is to determine whether the microbiota and biogenic molecules found in sea air are also found in the nasal swabs of the participants. In this way, the investigators will gain an understanding of which sea air components are inhaled by humans and how this changes over time.
2. Second, the investigators want to get an idea of whether these inhaled sea air components have an effect on certain pathways in the human body. In the in vitro study with cell lines, effects were already seen of sea air exposure on certain pathways in the body. Now the second goal of this study, is to see if changes in immunity biomarkers (IL-6, TNF-alpha, IL-10) are seen in vivo in humans. The Investigators will do this by taking VAMS blood samples from the participants.

ELIGIBILITY:
Inclusion Criteria:

* health participants between 18 and 50 years old

Exclusion Criteria:

* people with a medical condition
* people younger than 18 and older than 50

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
nose swabs: respiratory microbiome and biogenics profile | 4 times during the 8 week study period
  DNA from the nose swabs will be analysed for microbiota and biogenics on the swabs will be analysed as well, to get an idea of what molecules and microbiota from the sea air are inhaled.
VAMS blood samples: cytokines | 4 times during the 8 week study period
  Cytokines (IL-6, TNF-alfa, IL-10) will be measured in blood samples to link the sea air exposure to the human health

CONTACTS AND LOCATIONS:
Overall Officials: Hannelore Denys, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No